CLINICAL TRIAL: NCT06333470
Title: Liwan Eye Study: the Fourth Follow-up
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024KYPJ025
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Primary Angle-Closure Glaucoma
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Primary angle closure diseases — Primary angle-closure suspect (PACS), which is characterized by appositional angle closure, is the earliest stage of primary angle closure diseases and can finally progress to primary angle-closure glaucoma (PACG).

SUMMARY:
Primary angle-closure glaucoma (PACG) is one of the major causes of blindness affecting more than 20 million patients worldwide. The goals of this observational cohort study are to investigate the 20-year incidence of PACG in Chinese population aged 50 years and to develop prediction models for the long-term risk of progression from primary angle-closure suspect (PACS) to PACG.

DETAILED DESCRIPTION:
Primary angle-closure glaucoma (PACG) is potentially a devastating disease, responsible for half of glaucoma-related blindness worldwide, especially in East Asia. Primary angle-closure suspect (PACS), which is characterized by appositional angle closure, is the earliest stage of primary angle closure diseases and can finally progress to PACG. Thus, identifying PACS eyes at risk of angle closure is crucial for its management. However, the natural history of progression from PACS to PACG and its prediction models are still limited in long-term longitudinal studies. Meanwhile, visual impairment poses a significant global public health burden along with the accelerating trend of aging, it is imperative to further evaluate the visual impairment among the elderly population.

The Liwan Eye Study was a population-based study initiated in 2003. The decision to select Liwan District for the survey was taken because of its stable, older population and a socioeconomic profile representative of Guangzhou as a whole. At baseline, 1405 eligible subjects aged 50 years and older completed a comprehensive eye examination and a questionnaire interview regarding education, income, hypertension and diabetes mellitus. To improve the monitoring of PACS and prevent vision loss associated with PACG, the purposes of this observational cohort study are to investigate the 20-year incidence of PACG in Chinese population aged over 50 years, develop prediction models that include eye characteristics, demographic features, ocular imaging characteristics, and genetic factors for the long-term risk of progression from PACS to PACG. Moreover, we aim to investigate the 20-year change in visual impairment and associated factors.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have previously participated in the Liwan Eye Study
* Individuals who sign an informed consent form voluntarily

Exclusion Criteria:

* None

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All participants who will be follow-up in this study are from the Liwan Eye Study. At baseline, study subjects were enrolled in Liwan District, Guangzhou. (Liwan District is 1 of 10 administrative districts in Guangzhou, with a population of 514,600.) The decision to select this district for the survey was taken because of its stable, older population and a socioeconomic profile representative of Guangzhou as a whole. Individuals aged 50 years or more who had been resident in the selected study districts for more than 6 months were considered eligible during the enumeration. A total of 1405 eligible subjects were identified from the register.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The 20-year incidence of primary angle-closure glaucoma (PACG) in Chinese population aged over 50 years | 20-year
  The presence of PACG is determined by visual acuity, intraocular pressure, anterior segment optical coherence tomography (AS-OCT). The incidence of PACG is defined as the number of new cases of PACG divided by the number of individuals without PACG at baseline.

SECONDARY OUTCOMES:
The development of prediction models for the long-term risk of progression from primary angle-closure suspect (PACS) to primary angle-closure glaucoma (PACG) | 5-year, 10-year, 20-year
  Prediction model performance was assessed by discrimination and calibration.Discrimination was evaluated using the ROC curve and area under the curve (AUC) or C-statistics. Calibration was visualized through calibration plots and evaluated using the Hosmer-Lemeshow goodness-of-fit test (HL test).
The 20-year incidence of visual impairment in Chinese population aged over 50 years | 20-year
  Visual acuity (VA) will be measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR illiterate E VA chart. Visual impairment is defined as VA <20/60 & ≥20/400, and blindness is defined as VA<20/400 in the better-seeing eye.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: Yes
Available on request. The datasets generated from the current study will be available upon request from Dr Wei Wang (wangwei@gzzoc.com) after the study is completed.
Supporting Information: Study Protocol
Access Criteria: For access to the data, please contact the principal investigator after the study is completed.